CLINICAL TRIAL: NCT04689321
Title: Revision of the European Organisation for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire (QLQ)-BN20 Brain Tumour Module
Brief Title: Revision of the EORTC QLQ-BN20 Questionnaire
Acronym: QLQBN20
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Leiden University Medical Center (Other)
Collaborators: Medical Center Haaglanden (Other); Regina Elena Cancer Institute (Other); San Giovanni Addolorata Hospital (Other); NHS Lothian (Other Government); University Hospital Regensburg (Other); University Hospital, Bonn (Other); University of Zurich (Other); National Cancer Center, Japan (Other Government); King Hussein Cancer Center (Other); Clinical Hospital Center Rijeka (Other); Leeds Cancer Centre at St. James's University Hospital (Other)
Responsible Party: Principal Investigator, LindaDirven, Principal Investigator, Leiden University Medical Center
Other Study IDs: P18.095
Record Dates: First submitted 2020-12-22; First posted 2020-12-30 (Actual); Last update posted 2020-12-30 (Actual); Status verified 2020-12

CONDITIONS: Glioma; Brain Metastases, Adult
Keywords: health-related quality of life; patient-reported outcome; brain tumor
MeSH Terms: conditions — Glioma; Brain Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Phase 1: Patients recruited for phase 1 will undergo a semi-structured interview to identify issues that may be relevant to include in the revised EORTC QLQ-BN20 questionnaire.
  Interventions: Other: No intervention
- Phase 3: Patients recruited for phase 3 will complete the draft questionnaire, and rate each item for relevance, and indicate the 10 most important items. Also, a semi-structured interview will be conducted including debriefing questions to determine if the questionnaire is complete and the questions are acceptable.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — This is not an interventional study.

SUMMARY:
Despite the fact that use of the European Organisation for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire - Brain Neoplasm (QLQ-BN20) has tremendously contributed to insight into the health-related quality of life (HRQoL) of brain tumor patients, certain items of the questionnaire have raised issues, and new treatments have been introduced, with different toxicity profiles not covered by the current measure. These observations have led to the recognition that a revision of the QLQ-BN20 is warranted.

The aim of this project is to update the current EORTC QLQ-BN20 questionnaire.

DETAILED DESCRIPTION:
The European Organisation for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire - Brain Neoplasm (QLQ-BN20) brain tumor module was developed and validated in 1996, with a phase IV validation in 2010. The aim of this module was to evaluate the effects of the tumor and its treatment on symptoms, functions and health-related quality of life (HRQoL) of brain tumor patients, both in clinical trials and clinical practice.

An unpublished systematic review conducted by our group revealed that since the publication of the QLQ-BN20 in 1996, there has been an increase in the use of this questionnaire, not only in glioma patients for whom this questionnaire was developed, but also in meningioma patients, patients with brain metastases or groups with mixed types of brain tumors. The use of the QLQ-BN20 showed an increase over time: from 20 publications in the period 1996-2006, to 98 publications in the period 2007-2016.

One of the reasons for updating the current QLQ-BN20 questionnaire is that were have encountered limitations in the use of specific items. For example, the item referring to the occurrence of seizures results in an underestimation of the true prevalence of seizures. In previous clinical studies it was shown that 30-60% of the brain tumor patients experience seizures. In contrast, large randomized controlled trials using the QLQ-BN20 to determine seizure occurrence showed prevalences of only 6 to 14 percent. This is probably due to the time frame that is used for this item, i.e. the 'last week'. Although seizures are frequent, they often do not occur weekly. With the current response format, detection of seizures is difficult and this should be taken into account in the revision of the QLQ-BN20 questionnaire. Second, several items show severe floor-effects. Probably the most important reason to revise the current QLQ-BN20 questionnaire is because major advances in the treatment of brain tumors have been made in the last 20 years. Compared to 20 years ago, when the QLQ-BN20 was developed, current standard treatment (multimodal treatment including surgery, radiotherapy and chemotherapy) is different and treatments have a different toxicity profile. Moreover, new treatment opportunities are currently explored and include targeted treatment and immunotherapy. These types of treatment bring new toxicities, e.g. eye, skin and endocrine function problems. The current brain tumor module lacks sufficient coverage of domains that are affected by current and new treatment options.

Thus, despite the fact that use of the QLQ-BN20 has tremendously contributed to insight into the quality of life of brain tumor patients, several observations have led to the recognition that a revision of the QLQ-BN20 is warranted. Therefore, the aim of this project is to update the current EORTC QLQ-BN20 questionnaire.

Aim: The overall aim of this study is to update the current EORTC QLQ-BN20 questionnaire for use in brain tumor patients.

Study design: The methods for this prospective study will follow the EORTC Quality of Life Group guidelines for updating existing modules, including a literature review, interviews with patients and health care professionals (for the identification of items relevant to current/new treatments (phase I)), creation of a revised item list (phase II), and psychometric pilot testing (phase III).

Phase 1: Semi-structured interviews with 27 patients and 6 healthcare professionals to identify relevant issues for brain tumor patients (these issues are identified with a systematic literature review and have to reflect the patients' functioning and well-being, such as symptoms / impairments, activities in daily life and participation restrictions).

Phase 2: Construction of a comprehensive item list with items that are relevant for brain tumor patients (including construction of items, and translations).

Phase 3: The draft item list resulting from phase II will be pretested in 108 patients from at least 6 countries in 4 main European regions and Asia (Netherlands, Germany, Italy, United Kingdom, Switzerland, Croatia, Jordan and Japan). The primary aim of pretesting the module is to identify and solve potential problems (phrasing, sequence questions) and to identify missing or redundant items. Second, preliminary psychometric testing will be performed.

The questionnaire resulting from phase III will subsequently be field-tested in a large, international group of patients in order to determine its acceptability, reliability, validity, responsiveness and cross-cultural applicability. This is currently not part of the study protocol, but will commence after phase III is successfully completed.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven or suspected diffuse astrocytoma (Isocitrate Dehydrogenase-1 (IDH-1) wildtype or IDH-1 mutated), diffuse oligodendroglioma (IDH-1 mutated and 1p/19q co-deleted), anaplastic astrocytoma (IDH-1 wildtype or IDH-1 mutated), anaplastic oligodendroglioma (IDH-1 mutated and 1p/19q co-deleted), glioblastoma (IDH-1 wild-type or IDH-1 mutated), or diffuse astrocytoma not otherwise specified (NOS), anaplastic astrocytoma NOS, oligodendroglioma NOS, oligoastrocytoma NOS, anaplastic oligoastrocytoma NOS, anaplastic oligodendroglioma NOS or glioblastoma NOS; or radiologically verified metastatic brain tumour.
* Adult patients: ≥18 years of age
* Willing to provide written informed consent

Exclusion Criteria:

* Patients without understanding of the official language of the country in which they live.
* Patients with any psychiatric condition or cognitive impairment, as determined by the treating physician, that would hamper undergoing semi-structured interviews.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of both patients with a primary brain tumor (histologically confirmed glioma) and metastatic brain tumor (brain metastases with a histologically confirmed primary tumor) who visit the outpatient clinic in The Netherlands, United Kingdom, Italy, Germany, Poland or Japan.
Sampling Method: Non-Probability Sample
Enrollment: 135 (Estimated)
Dates: Start 2018-12-19 (Actual); Primary Completion 2024-01-01 (Estimated); Study Completion 2024-01-01 (Estimated)

PRIMARY OUTCOMES:
Number of relevant items of the EORTC QLQ-BN101 | Baseline
  Construction of the final item list, based on predefined decision rules

SECONDARY OUTCOMES:
Number of multi-item and single-item scales | Baseline
  Exploratory Factor Analysis to determine multi-item and single-item scales (scales not yet known; items are scored on a 4-point Likert scale ranging from 'Not at all' to 'Very much')
Internal consistency | Baseline
  The internal consistency of the scales will be explored using Cronbach's alpha (scales not yet known; response options for each item are based on a 4-point Likert scale ranging from 'Not at all' to 'Very much')
Convergent validity | Baseline
  Convergent validity of the final item list will be assessed by means of inter-item correlations
Discriminant validity | Baseline
  Discriminant validity of the final item list will be assessed by means of known-group comparisons

CONTACTS AND LOCATIONS:
Overall Officials: Linda Dirven, PhD, Principal Investigator — Leiden University Medical Center
Locations (1):
- Leiden University Medical Center, Leiden, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No
This study is funded by the European Organisation for Research and Treatment of Cancer, and data will be stored there. Researchers can request data according to the EORTC's data sharing policy.